CLINICAL TRIAL: NCT00526799
Title: A Phase I/II Study of Sorafenib in Combination With Topotecan for the Treatment of Platinum-Resistant Recurrent Ovarian Cancer or Primary Peritoneal Carcinomatosis: Hoosier Oncology Group GYN06-111
Brief Title: Sorafenib + Topotecan for Platinum-Resistant Recurrent Ovarian Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed to accrual due unfavorable interim analysis
Sponsor: Daniela Matei, MD (Other)
Collaborators: Bayer (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Daniela Matei, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN06-111
Record Dates: First submitted 2007-09-05; First posted 2007-09-10 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sorafenib; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Experimental): Topotecan 3.5 mg/m^2 + Sorafenib dose escalation:
  Interventions: Drug: Sorafenib; Drug: Topotecan
- Phase II (Experimental): Topotecan 3.5 mg/m^2 + Sorafenib 400 mg po daily.
  Interventions: Drug: Sorafenib; Drug: Topotecan

INTERVENTIONS:
Drug: Sorafenib — Phase I: Dose Escalation, Phase II: MTD
  Dose level -1: 200mg po daily Dose level 1: 400mg po daily (MTD) Dose level 2: 400mg po bid
Drug: Topotecan — 3.5mg/m2 weekly, 3 weeks on and one week off.

SUMMARY:
This multi-institutional phase I/II clinical trial will test the tolerability and efficacy of the combination sorafenib and topotecan in patients with recurrent ovarian cancer, which is platinum-resistant (recurrence within 6 months from completing platinum based therapy) or refractory (progressive disease during platinum based therapy).

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Topotecan: 4mg/m2 weekly, 3 weeks on and one week off.
* Sorafenib: Assigned cohort dose for phase I (up to 12 patients) Maximum tolerated dose for phase II (21 total patients)

Cycles will consist of 4 weeks (28 days) with disease evaluations every 8 weeks.

Non-PD and acceptable toxicity: Patients will continue protocol therapy PD or unacceptable toxicity: Patients will discontinue protocol therapy

ECOG performance status 0-1

Life expectancy: Three (3) months

Hematopoietic:

* White blood cell count (WBC) > 3 K/mm3
* Hemoglobin (Hgb) > 9 g/dL
* Platelets > 100 K/mm3
* Absolute neutrophil count (ANC) > 1.5 K/mm3
* INR < 1.5 or a PTT within normal limits. NOTE: Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate.
* No evidence or history of bleeding diathesis or coagulopathy.

Hepatic:

* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST, SGOT) < 2.5 x ULN
* Alanine aminotransferase (ALT, SGPT) < 2.5 x ULN
* Alkaline phosphate < 2.5 x ULN

Renal:

* Creatinine < 1.5 x ULN

Cardiovascular:

* No history of myocardial infarction or angina pectoris or angina equivalent within 6 months prior to registration for protocol therapy (the patient may not be on anti-anginal or anti-arrhythmic medications), or have uncontrolled hypertension or congestive heart failure > class II NYHA

Pulmonary:

* No thrombolic or embolic events such as a cerebrovascular accident, including transient ischemic attacks within the past 6 months.
* No pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 28 days prior to registration for protocol therapy.
* No non-pulmonary hemorrhage/bleeding event > CTCAE Grade 3 within 28 days prior to registration for protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically-confirmed epithelial ovarian cancer, primary peritoneal carcinomatosis or fallopian tube cancer. Enrollment of patients with clear cell histology is encouraged.
* Have measurable disease according to RECIST or detectable disease by 1) CA-125 at least twice the ULN within 14 days prior to registration for protocol therapy; 2) Ascites and/or pleural effusion attributed to tumor; 3) solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST definitions for target lesions.
* Have failed at least one prior platinum based chemotherapeutic regimen.
* No more than 3 prior treatment regimens for epithelial ovarian cancer.
* Prior radiation therapy is allowed to < 25% of the bone marrow.
* Be at least 4 weeks since last anti-cancer treatment, radiation or surgery at the time of registration for protocol therapy.
* No active cancer in addition to the epithelial ovarian cancer within the last 5 years, with the exception of: superficial skin cancer (basal cell or squamous cell skin carcinoma; carcinoma in situ of the cervix; Stage I endometrial cancer with less than 50% invasion of the myometrium, or other adequately treated Stage I or II cancer in complete remission.
* Age > 18 years at the time of consent
* Written informed consent and HIPAA authorization for release of personal health information.
* Females of childbearing potential must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 90 days after treatment discontinuation
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.

Exclusion Criteria:

* No known or suspected allergy to sorafenib or any agent given in the course of this trial.
* No prior treatment with anti-angiogenesis therapy.
* No active CNS metastases.
* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
* No concurrent combination anti-retroviral therapy for the treatment of immunodeficiency.
* No clinically significant infections requiring antibiotic treatment.
* No evidence of bowel obstruction, malabsorption, or other contraindication to oral medication.
* No serious non-healing wound, ulcer, or bone fracture.
* No major surgery, open biopsy or significant traumatic injury within 28 days of registration for protocol therapy.
* No use of St. John's Wort or rifampin (rifampicin) while on protocol therapy.
* No condition that impairs patient's ability to swallow whole pills.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, M.D., Study Chair — Hoosier Oncology Group, Inc.
Locations (8):
- United States (8):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Hospital Cynecologic Oncology, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Schwartz Gynecologic Oncology, PLLC, Brightwaters, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matei D, Emerson RE, Schilder J, Menning N, Baldridge LA, Johnson CS, Breen T, McClean J, Stephens D, Whalen C, Sutton G. Imatinib mesylate in combination with docetaxel for the treatment of patients with advanced, platinum-resistant ovarian cancer and primary peritoneal carcinomatosis : a Hoosier Oncology Group trial. Cancer. 2008 Aug 15;113(4):723-32. doi: 10.1002/cncr.23605. PMID 18618737
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Topotecan 3.5 mg/m^2 + Sorafenib assigned dose level:
  Sorafenib Dose level -1=200 mg po daily Sorafenib Dose level 1=400 mg po daily Sorafenib Dose level 2=400 mag po bid
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 16 | 14
Completed | 15 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Intercurrent Complicating Disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Median (Full Range); unit: years] | 52.5 [41 to 66] | 52.5 [35 to 79] | 52.5 [35 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Eastern Cooperative Onocology Group (ECOG) Perfomance Status [Number; unit: participants] — ECOG: Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead
  participants
    ECOG=0 | 9 | 13 | 22
    ECOG=1 | 7 | 1 | 8
Origin of Cancer [Number; unit: participants]
  Epithelial Ovarian Cancer | 14 | 13 | 27
  Primary Peritoneal Carcinomatosis | 2 | 1 | 3
Histology [Number; unit: participants]
  Serous Papillary | 8 | 12 | 20
  Clear Cell | 1 | 0 | 1
  Endometroid | 4 | 1 | 5
  Other | 3 | 1 | 4
Number of Prior Therapies [Median (Full Range); unit: Prior Therapies] | 2 [1 to 3] | 3 [1 to 3] | 2 [1 to 3]
Response Evaluation [Number; unit: participants] — Response Evaluation Criteria in Solid Tumors (RECIST):
  Measurable disease is defined by the presence of at least one measureable lesion. If the measureable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology.
  Detectable disease is defined as a patient who does not have measureable disease, but has at least one: 1)CA-125 >= 2x ULN w/in 14d prior to registration 2)Ascites and/or pleural effusion attributed to tumor; 3)solid and/or cystic abnormalities on radiographic imaging that don't meet RECIST definitions for target lesions.
  participants
    Measurable Disease (RECIST) | 10 | 12 | 22
    Detectable Disease | 6 | 2 | 8
Platinum Sensitivity [Number; unit: participants]
  Platinum refractory | 5 | 4 | 9
  Platinum Resistant | 10 | 8 | 18
  Platinum allergy | 1 | 2 | 3
CA125 at Enrollment [Median (Full Range); unit: U/mL] | 744.2 [144.7 to 2771.5] | 1669.0 [437.0 to 2901.0] | 744.2 [144.7 to 2901.0]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: An initial 3 patients will be enrolled at dose level 1. If all 3 patients in dose level 1 complete the first cycle of therapy without a dose limiting toxicity (DLT), 3 patients will be enrolled at dose level 2. If 0 of 3 or 1 of 6 patients in dose level 2 experience a DLT, all subsequent patients will be enrolled in the Phase II cohort at dose level 2. If 2 of the first 3 or 2 of the total 6 patients experience DLT at dose level 2, then dose level 1 will be considered the MTD and used in the second phase.
Time Frame: Each participant was treated at their assigned dose level on 28 day cycles until disease progression or unacceptable toxicity. Participants were evaluated for toxicity every two weeks.
Population: Of the 16 patients enrolled in the phase I study, five were not evaluable for MTD determination due to intercurrent illnesses interfering with toxicity assessment or withdrawal and were replaced or excluded.
Measure: Number; unit: mg/day
Groups:
- Phase I Participants: Phase I Participants evaluable for MTD
Arm/Group | Phase I Participants
Number analyzed (Participants) | 11
mg/day | 400

2. Primary Outcome: Percentage of Participants With Response
Description: To assess response in patients with recurrent or resistant epithelial ovarian cancer treated with Sorafenib plus Topotecan. Reponse evaluated per RECIST criteria where:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Disease assessments were conducted on the 8th week (Cycle 2, Week 4) and every eight weeks there after, until treatment discontinuation
Measure: Number; unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 14
percentage of participants
  partial reponse | 7.1
  stable disease | 71.4
  progressive disease | 14.3
  unevaluable | 7.1
  complete response | 0

3. Secondary Outcome: Progression-free Survival
Description: To determine the progression-free survival of patients treated with Sorafenib plus Topotecan.
Time Frame: From enrollment until treatment discontinuation. Participants may remain on study drug indefinitely
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase I & II: Topotecan 3.5 mg/m^2 + Sorafenib 400 mg po daily during phase II.
  During phase I:
  Topotecan 3.5 mg/m^2 + Sorafenib assigned dose level:
  Sorafenib Dose level -1=200 mg po daily Sorafenib Dose level 1=400 mg po daily Sorafenib Dose level 2=400 mag po bid
Arm/Group | Phase I & II
Number analyzed (Participants) | 30
months | 3.7 [3.0 to 5.5]

4. Secondary Outcome: Clinical Benefit
Description: To determine the rate of clinical benefit defined as the percentage of patients experiencing an objective response or a CA125 response.
Time Frame: From enrollment until treatment discontinuation. Participants may remain on study drug indefinitely
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Phase II
Number analyzed (Participants) | 14
percentage of particpants | 71.4 [41.9 to 91.6]

5. Secondary Outcome: Duration of Stable Disease
Description: To determine duration of stable disease, in months
Time Frame: From enrollment until treatment discontinuation. Participants may remain on study drug indefinitely
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 14
months | 4.2 [3.4 to 5.5]

ADVERSE EVENTS:
Time Frame: Duration of Study
Description: Combined Phase I/Phase II safety data
Groups:
- Phase I/Phase II: All Phase I/Phase II participants
Arm/Group | Phase I/Phase II
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/Phase II (N=30)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OBSTRUCTION, GI / SMALL BOWEL NOS (Gastrointestinal disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/Phase II (N=30)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 3 (5)
ALKALINE PHOSPHATASE (Investigations) | 5 (5)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 2 (2)
ANOREXIA (Gastrointestinal disorders) | 6 (14)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 1 (1)
ASCITES (NON-MALIGNANT) (Gastrointestinal disorders) | 2 (10)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 4 (4)
AUDITORY/EAR - OTHER (SPECIFY, __) (Ear and labyrinth disorders) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 5 (8)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 17 (21)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CREATININE (Investigations) | 2 (3)
DEHYDRATION (Gastrointestinal disorders) | 3 (8)
DENTAL: DENTURES OR PROSTHESIS (Gastrointestinal disorders) | 1 (1)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 7 (12)
DIZZINESS (Nervous system disorders) | 1 (1)
DRY EYE SYNDROME (Eye disorders) | 1 (1)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 9 (9)
EDEMA: LIMB (Blood and lymphatic system disorders) | 3 (3)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 16 (31)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (1)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 1 (1)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 5 (7)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 5 (7)
HEMOGLOBIN (Blood and lymphatic system disorders) | 17 (43)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHAGE/BLEEDING - OTHER (SPECIFY, __) (General disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / BRONCHUS (Infections and infestations) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / UPPER AIRWAY NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / EXTERNAL EAR (OTITIS EXTERNA) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SOFT TISSUE NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 12 (19)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 9 (17)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 4 (6)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 5 (6)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 3 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 4 (7)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 1 (2)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 19 (39)
NEUROPATHY: MOTOR (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 12 (12)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 15 (42)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 13 (16)
PAIN / BACK (General disorders) | 5 (6)
PAIN / BLADDER (Renal and urinary disorders) | 1 (1)
PAIN / BREAST (Reproductive system and breast disorders) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 4 (10)
PAIN / FACE (General disorders) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 2 (2)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 4 (4)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / ORAL CAVITY (Gastrointestinal disorders) | 1 (1)
PAIN / PAIN NOS (General disorders) | 1 (1)
PAIN / PELVIS (General disorders) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 1 (2)
PHOSPHATE, SERUM-LOW (HYPOPHOSPHATEMIA) (Investigations) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 12 (38)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 4 (6)
PROTEINURIA (Investigations) | 2 (2)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 5 (5)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 1 (2)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 6 (6)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 5 (5)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 2 (2)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 1 (1)
URTICARIA (HIVES, WELTS, WHEALS) (Skin and subcutaneous tissue disorders) | 1 (3)
VOMITING (Gastrointestinal disorders) | 9 (20)
WEIGHT LOSS (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No